CLINICAL TRIAL: NCT04950647
Title: Efficacy and Safety of Nitrazine in the Treatment of Amyotrophic Lateral Sclerosis: a Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Study
Brief Title: Efficacy and Safety of Nitrazine in the Treatment of ALS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: West China Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D2020109
Record Dates: First submitted 2021-06-27; First posted 2021-07-06 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-06

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test group 1 (Experimental): Nitroketazine tablet 600 mg group
  Interventions: Drug: Nitrofurazone Group 1
- Test group 2 (Experimental): Nitroketazine tablets 1200 mg group
  Interventions: Drug: Nitroketazine Group 2
- Control group (Placebo Comparator): placebo group
  Interventions: Drug: placebo group

INTERVENTIONS:
Drug: Nitrofurazone Group 1 — Test group 1: Nitroketazine tablet 600 mg group (Nitroketazine 300 mg tablet X2 + placebo 300 mg tablet ×2 tablets each time; If the subject progresses and cannot take 300mg tablets, Nitroketazine 100mg tablets x6 + placebo 100mg tablets x6) can be replaced.
  Arms: Test group 1
Drug: Nitroketazine Group 2 — Test group 2: Nitroketazine tablets 1200 mg group (each oral Nitroketazine 300 mg tablets x4 tablets; If the subject progresses and cannot take 300 mg tablets, Nitroketazine 100mg tablets x12 tablets can be taken instead).
  Arms: Test group 2
Drug: placebo group — Control group: placebo group (placebo 300mg tablets x4 tablets each orally; If subjects progress and cannot take 300mg tablets, they may take placebo 100 mg tablets x 12 tablets instead).
  Arms: Control group

SUMMARY:
To evaluate the trend of safety and effectiveness of Nitroketazine tablets for ALS patients, and to explore the best effective dose.

DETAILED DESCRIPTION:
This trial was a randomized, double-blind, placebo-controlled parallel design. Patients with ALS were selected by inclusion exclusion criteria, and then randomly assigned to receive either the experimental drug or placebo. Test group 1: Nitroketazine tablet 600mg group (Nitroketazine 300mg tablet x2 + placebo 300mg tablet x2 each time; If the subject progresses and cannot take 300 mg tablets, Nitroketazine 100mg tablets x6 tablets + placebo 100mg tablets x6 tablets can be taken instead). Test group 2: Nitroketazine tablets 1200 mg group (each oral Nitroketazine 300 mg tablets x4 tablets; If the subject progresses and cannot take 300 mg tablets, Nitroketazine 100 mg tablets x12 tablets can be taken instead). Control group: placebo group (placebo 300mg tablets x4 tablets each orally; If subjects progress and cannot take 300 mg tablets, they may take placebo 100mg tablets x 12 tablets instead). Usage: Oral administration, twice a day, once in the morning and once in the evening (or the interval between two medication is 28h), at least 1" hour before meal (21 h before meal) on an empty stomach or at least 2 hours after meal (22h after meal) on an empty stomach, 180±3 days. Eligible subjects will start treatment on Day 1 after randomization, and visit the study center at the end of 1, 3, and 6 (or when they quit the study midway) for safety and efficacy checks. Telephone interviews were conducted at the end of the seventh day of treatment, the end of the second month, the end of the fourth month, the end of the fifth month of treatment, and the second week after the end of the sixth month of treatment. A total of 150 ALS patients were planned to be enrolled, with 50 patients in each group.

ELIGIBILITY:
Inclusion Criteria:

1. Age 45-70, gender unlimited (including 45 and 70);
2. diagnoses in accordance with the confirmed and proposed ALS diagnostic standards ofthe Revised World Federation of Neurology (1998);
3. The duration of disease from onset to randomization of subjects is less than 2 years;
4. Before randomization, ALSFRS-R scores were ≥2 points, and respiratory function items were 4 points;
5. ALSFRS-R decreased by 1-4 points in screening period 3A (≥1 and lt; 4);
6. Random pre-respiratory function Forced Vital Capacity (%FVC) ≥80%;
7. Understand and abide by the test procedures, participate voluntarily, and sign the informed consent (the informed consent should be signed by the person or the guardian voluntarily).

Exclusion Criteria:

1. Familial ALS (judged by family history);
2. Patients with significant cognitive impairment (MMSE: illiteracy group < 19 points, elementary school. 22 points, S26 points in the junior high school and above group (more than 8 years of education);
3. obvious dysphagia;
4. Severe renal insufficiency: creatinine clearance. 30 mL/min (Cockcroft-Gault formula), or other known severe renal insufficiency;
5. Severe liver function impairment: ALT, AST&GT; 3 times the upper limit of normal value, or other known liver diseases such as acute or chronic active hepatitis, cirrhosis, etc.;
6. In the screening stage, patients with heart failure who developed acute myocardial infarction or underwent interventional therapy within the last 6 months (grade II1-IV according to NYHA);
7. Complicated with malignant tumors, serious diseases of blood, digestion or other systems.
8. Allergic to experimental drugs or ligustrazine;
9. Pregnancy and lactation;
10. Participated in, or is participating in, other clinical trials within 30 days prior to screening;
11. The investigator did not consider it appropriate to participate in this study.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
ALSFRS-R score | Treatment day 180
  ALSFRS -r score difference between the difference in value relative to the baseline group;

SECONDARY OUTCOMES:
grip strength | Treatment day 180
  Intergroup differences in grip strength relative to baseline difference

CONTACTS AND LOCATIONS:
Overall Officials: Dongsheng Fan, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes